CLINICAL TRIAL: NCT02416154
Title: IFN-epsilon and Hormonal Contraceptive Modulation of the Risk of HIV Acquisition, Part 1: Expression in the Female Reproductive Tract
Brief Title: Expression of IFN-epsilon in the Female Reproductive Tract
Acronym: Epsilon
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); MIMR-PHI Institute, Australia (Unknown)
Responsible Party: Principal Investigator, Sharon Achilles, Assistant Professor, University of Pittsburgh
Other Study IDs: OPP1108501
Record Dates: First submitted 2015-04-09; First posted 2015-04-14 (Estimated); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Interferon Expression in the Female Reproductive Tract
Keywords: interferon-epsilon; female reproductive tract; neopterin; menstrual cycle
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — whole blood plasma vaginal swabs cervical swabs Vaginal fluid collected by sponge cervicovaginal lavage fluid cervical cells collected by cytobrush vaginal biopsies cervical biopsies endometrial biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Follicular phase: Normally cycling women in the follicular phase of menses
  Interventions: Procedure: Reproductive tract and blood sampling
- Luteal phase: Normally cycling women in the luteal phase of menses
  Interventions: Procedure: Reproductive tract and blood sampling

INTERVENTIONS:
Procedure: Reproductive tract and blood sampling — Reproductive tract and blood sampling will be performed at enrollment only in this cross-sectional parallel cohort study.

SUMMARY:
The proposed study aims to determine the expression of Interferon-ε (IFNε) in the female genital tract, which has never been mapped before in humans. High expression in other mammalian female reproductive tract (FRT) has been suggested to be important in anti-sexually transmitted infection (STI)/HIV immunity and its expression decreases with progestogen treatment. Future studies are planned to understand if hormonal contraceptives affect the presence of interferon in the healthy female genital tract, potentially changing the risk of for STI and HIV.

DETAILED DESCRIPTION:
Objectives:

1. To optimize measurement protocols for IFNε and related biomarkers in samples from the female reproductive tract.
2. To quantify and characterize IFNε expression in the upper and lower genital tract and blood in normally cycling women during the follicular and luteal phases of the menstrual cycle.

Study design: This is a single site, parallel cross-sectional study

Specific Aims:

The aim of this study is to determine which "IFNε -related assays" can be performed on different types of FRT samples. The possible "IFNε-related assays" are:

* IFNε messenger ribonucleic acid (mRNA) levels by quantitative reverse transcriptase polymerase chain reaction (qRT PCR) (requiring frozen tissue processed for RNA)
* IFN Regulated Gene expression by qRT PCR, microarray or targeted gene set using Fluidigm platform (frozen tissue)
* PR and ER gene expression (as above)
* IFNε tissue protein levels* (by immunoassay) and progesterone and estrogen receptors (PR/ER) by Western blotting (frozen tissue)
* IFNε and Neopterin (a well characterized compound whose production can be stimulated by IFNs and whose specificity in this setting needs validation) or other IFNε-biomarkers** by immunoassay in cervicovaginal lavage (CVL) fluids
* Immunohistochemistry of IFNε, PR/ER, + other (e.g. cells, cytokines) (fixed tissue)

  * Studies of FRT samples from wild type and IFNε-/- mice would be used to first validate Neopterin as a "biomarker" of IFNε activity in the FRT; and microarray analyses may reveal other secreted proteins that may be used as "biomarkers" of IFNε activity.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 through 35 years (inclusive) at screening
2. Non-pregnant women in general good health as determined by the site clinician
3. Premenopausal with history of regular menstrual cycles (regular cycles defined as occurring every 21-35 days when not using hormones and with a variation of typical cycle length of no more than 5 days)
4. Regular and consistent condom use, prior surgical sterilization by participant or sexual partner, or heterosexually abstinent since last menses prior to enrollment
5. Able and willing to provide written informed consent to be screened for and to take part in the study, including willingness to undergo all study-related assessments and follow all study-related procedures
6. Able and willing to provide adequate locator information
7. HIV-uninfected based on testing performed by study staff at enrollment

Exclusion Criteria:

1. Use of any hormonal or intrauterine contraceptive method within 30 days of enrollment
2. Use of depot medroxyprogesterone acetate (DMPA) within 10 months of enrollment
3. Pregnancy or breastfeeding within 60 days of enrollment
4. Surgical procedure involving the pelvis in the 30 days prior to enrollment (includes dilation and curettage, cryosurgery and biopsy of the vagina, vulva, cervix, and endometrium)
5. Internal vaginal use of any device (includes sex toys, cervical caps, diaphragms, menstrual collection devices, and pessaries; excludes tampons and condoms) or product (includes spermicide, microbicide, douche, antifungal, steroid, or hormone) in the 30 days prior to enrolment (includes investigational products and devices)
6. New sexual partner within 90 days of enrollment
7. Urogenital infection or suspected infection within 30 days of enrollment including: symptomatic candidiasis, trichomonas vaginalis, and symptomatic bacterial vaginosis; or cervical infection, including N. gonorrhoea (GC), C. trachomatis (CT), or mucopurulent cervicitis; syphilis; herpes simplex virus (HSV) lesions, or other sores (Note: seropositive HSV without active lesions will not be excluded); acute pelvic inflammatory disease; urinary tract infection; recent exposure to a partner with GC, CT, Trichomonas, syphilis, or non-gonococcal urethritis (NGU)
8. Any history of immunosuppression (includes diabetes, HIV infection, and chronic steroid use or other immunosuppressive medications)
9. Antibiotic or antifungal therapy (vaginal or systemic) within 30 days of enrollment
10. Menses or other vaginal bleeding at the time of enrollment* (*Women who have vaginal bleeding at the scheduled enrollment visit may return at a different date to be re-examined and possibly enrolled provided they are still within the 90-day screening window and meet all criteria).
11. Vaginal or anal intercourse within 36 hours prior to enrollment
12. Heterosexual intercourse since last menses that places the participant at risk of pregnancy (without condom use or sterilization of at least one partner)
13. History of hysterectomy
14. History of malignancy within the pelvis (includes uterus, cervix, vagina, and vulva)
15. Any condition that, in the opinion of the Investigator, would preclude provision of consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy females aged18 through 35 years (inclusive) at screening
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Interferon epsilon expression | baseline
  Interferon epsilon expression will be assessed in the female reproductive tract and blood in women in the follicular phase of menses vs the luteal phase of menses in this cross-sectional study.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hertzog, PhD, Principal Investigator — Hudson Institute of Medical Research
Locations (2):
- United States (2):
  - Center for Family Planning Research, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania